CLINICAL TRIAL: NCT03272126
Title: Importance of Dosing Regimen for the Effect of Vitamin D Supplementation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TromsøEndo-2017-1
Record Dates: First submitted 2017-06-15; First posted 2017-09-05 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2017-09

CONDITIONS: Hypovitaminosis D
Keywords: vitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vitamin D bolus (Experimental): vitamin D 160 000 IU given as bolus
  Interventions: Drug: Vitamin D
- vitamin D daily (Experimental): vitamin D 4000 IU daily for 28 days
  Interventions: Drug: Vitamin D
- placebo (Placebo Comparator): identical looking as vitamin d
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — vitamin D given as bolus versus daily dosing
  Arms: vitamin D bolus; vitamin D daily
Drug: Placebo — identical looking as vitamin D
  Arms: placebo

SUMMARY:
Vitamin D is a hormone with effects not only on the skeleton, but on most tissues in the body. Lack of vitamin D is associated with cardio-vascular disease (CVD), type 2 diabetes, cancer, infectious and immunological diseases, as well as risk factors for these diseases. However, intervention studies with vitamin D have been inconclusive regarding diseases and risk factors. This could be due to inclusion of subjects already vitamin D sufficient, and short and underpowered studies. In addition, there are indications that the dosing regimens may be important, so that daily doses with vitamin D are more efficient than intermittent doses, which so far have been generally used. This could be related to the concentration of circulating and thereby intracellular vitamin D concentrations, which probably is dependent on daily vitamin D doses. This will be tested in the present study where 60 subjects will be randomized to vitamin D 160 000 once, vitamin D 4000 IU/day, or placebo for four weeks. The primary endpoints will be effects on serum hepcidin and plasma cathelicidin after 4 weeks, with effects on serum PTH, RNA expression and microRNA in peripheral blood, telomerase activity in peripheral blood mononuclear cells and the ration between serum 1,25(OH)2D and 24,25(OH)2D as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:- Males and females 20 - 70 years

* 20 kg/m2 > BMI < 35 kg/m2
* systolic BP < 175 mmHg, diastolic BP < 105 mmHg
* Serum 25(OH)D level < 50 nmol/L. Serum 25(OH)D < 50 nmol/L is considered as vitamin D deficiency, and accordingly, effects of vitamin D supplementation will be easier to detect than if the included subjects were vitamin D sufficient.
* Hgb, SR, CRP, creatinine < 130 umol/L in males, < 120 umol/L in females, calcium, FT4 and TSH within the normal reference range; ASAT < 90 mU/L ALAT < 140 U/L, HbA1c < 6.6 %
* The subjects must agree not to take any vitamin D supplementation, including cod liver oil or "mølje", use solarium or go on sunny vacation during the intervention period.

Exclusion Criteria:

* subjects allergic to peanuts
* subjects with primary hyperparathyroidism
* granulomatous diseases (sarcoidosis, tuberculosis, Wegner's granulomatosis)
* diabetes
* renal stones the last five years
* subjects seriously ill (or with chronic disease) and unfit for participation in the study (as judged by one of the study doctors)
* subjects using vitamin D supplements exceeding 800 IU per day or active vitamin D drugs (Rocaltrol or Etalpha)
* pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Hepcidin change | 4 weeks
  Difference between vitamin D given as a bolus 160 000IU vs 4000 IU regarding change in serum hepcidin

SECONDARY OUTCOMES:
Difference in serum PTH after 1 month | 4 weeks
  Difference between vitamin D given as a bolus 160 000IU vs 4000 IU regarding change in serum PTH, cathelicidin, RNA expression and micro RNA in peripheral blood, telomerase activity and the ratio between 1,25(OH)2D and 24,25(OH)2D, after 1 month
Difference in micro RNA Expression after 1 month | 4 weeks
  Difference between vitamin D given as a bolus 160 000IU vs 4000 IU
Difference in serum cathelicidin after 1 month | 4 weeks
  Difference between vitamin D given as a bolus 160 000IU vs 4000 IU
Difference in RNA Expression after 1 month | 4 weeks
  Difference between vitamin D given as a bolus 160 000IU vs 4000 IU
Difference in telomerase Activity after 1 month | 4 weeks
  Difference between vitamin D given as a bolus 160 000IU vs 4000 IU
Difference in ratio between 1,24(OH)2D and 24,24(OH)2D after 1 month | 4 weeks
  Difference between vitamin D given as a bolus 160 000IU vs 4000 IU

CONTACTS AND LOCATIONS:
Overall Officials: rolf jorde, MD PhD, Principal Investigator — UiT, Tromsø
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No